CLINICAL TRIAL: NCT07311668
Title: Accuracy of an Artificial Intelligence-Based System for Diagnosing Depressive Disorders: A Paired Comparison With Psychiatrist Clinical Diagnoses
Brief Title: Validation of the Accuracy of an AI-Based System for Diagnosing Depressive Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: MZhao-023
Record Dates: First submitted 2025-11-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-08

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The trial aimed to evaluate the accuracy of an artificial intelligence-based system for diagnosing depressive disorders. Specifically, it sought to determine whether the system's assessment validity is non-inferior to that of psychiatric specialists.

DETAILED DESCRIPTION:
This study evaluates the performance of the AI-assisted diagnostic system for identifying depressive disorders and its applicability in clinical settings. Utilizing a paired design with psychiatrists' clinical diagnoses as the gold standard, the study compares the system's diagnostic results with those of physicians to determine sensitivity and specificity, thus validating its clinical effectiveness in real-world outpatient scenarios. Additionally, standardized scales are used to assess users' perceptions of the system's usability, trustworthiness, and satisfaction, offering evidence to support the clinical integration of AI technology in mental health screening.

ELIGIBILITY:
1. Subjects with anxiety disorders （1）Inclusion Criteria:

   * In accordance with ICD-11 for Depressive Disorders;
   * Between the ages of 18-60;
   * Ability to use computers or smartphone;
   * Native Chinese speaker;
   * Signing informed consent. （2）Exclusion Criteria:
   * With severe psychiatric symptoms requiring hospitalization, or unable to complete the required assessment and treatment;
   * With a high risk of suicide or self-injury;
   * With severe physical diseases, central nervous system diseases, or substance abuse;
   * With intellectual, visual, or auditory impairments that affect their ability to interact with aided-diagnostic systems.
2. Health Control （1）Inclusion Criteria:

   * Not meet ICD-11 criteria for Mental Disorders;
   * Between the ages of 18-60;
   * Ability to use computers or smartphone;
   * Native Chinese speaker;
   * Signing informed consent. （2）Exclusion Criteria:
   * With mental illness, or unable to complete the required assessment and treatment;
   * With severe physical diseases, central nervous system diseases, or substance abuse;
   * With intellectual, visual, or auditory impairments that affect their ability to interact with aided-diagnostic systems.
3. Psychiatrist （1）Inclusion Criteria:

   * Over 18 years old;
   * A minimum of three years' experience in anxiety and other mental health fields;
   * Intermediate or higher professional title;
   * Currently employed in the selected test region;
   * Signing informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study includes the subjects with depressive disorders and healthy control into the experiment. Depressive individuals for the study will be recruited from actual outpatient patients at the Shanghai Mental Health Center. The healthy control will be recruited through public advertisements, both online and offline. Psychiatrists will be recruited through public advertisements by the Shanghai Mental Health Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy (Sensitivity, Specificity, and Area Under the Curve) of the AI-Based Screening System for Depressive Disorders | through study completion, an average of 1 week
  In this study, the evaluation results of the subjects were taken as the gold standard based on the diagnostic conclusions of psychiatrists. The screening results of the aided-diagnostic system were compared with the diagnostic conclusions of the psychiatrists to verify the screening effectiveness of this system. Sensitivity : Calculated as [True Positives / (True Positives + False Negatives)], evaluating the AI system's ability to correctly identify patients with depression. Specificity : Calculated as [True Negatives / (True Negatives + False Positives)], evaluating the AI system's ability to correctly exclude non-depressed individuals.Area Under the Receiver Operating Characteristic Curve (AUC), which comprehensively evaluates the diagnostic discriminative power of the system by plotting sensitivity versus 1-specificity across different decision thresholds and calculating the AUC value .

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No